CLINICAL TRIAL: NCT03405597
Title: HBsAb Response After HBV Vaccination in Chronic Hepatitis B Patients Who Have Lost HBsAg
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13/2560(EC1)
Record Dates: First submitted 2018-01-04; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Chronic Hepatitis B, HBsAg, Hepatitis B Vaccine
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Engerix-B

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy control (Experimental): Commercial Hepatitis B vaccine
  Interventions: Drug: Commercial Hepatitis B vaccine
- Chronic hepatitis B with vaccination (Experimental): Commercial Hepatitis B vaccine
  Interventions: Drug: Commercial Hepatitis B vaccine; Other: Standard Treatment
- Chronic hepatitis B without vaccination (Active Comparator): Standard treatment
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Drug: Commercial Hepatitis B vaccine — Commercial Hepatitis B vaccine (Engerix B) 20 microgram subcutaneous injection at month 0, 1, 6
  Other Names: Engerix B
  Arms: Chronic hepatitis B with vaccination; Healthy control
Other: Standard Treatment — HBsAg, HBsAb test Ultrasound upper abdomen every 6 months
  Arms: Chronic hepatitis B with vaccination; Chronic hepatitis B without vaccination

SUMMARY:
Chronic HBV infection is major problem in Asian countries. Years after chronic infection, in some cases serum HBsAg level declines to unmeasurable level. Some of patients develop anti-HBsAb but there is no standard treatment to accelerate HBsAg seroconversion.

There is a study to determine efficacy and safety of HBV vaccine in who is Chronic HBV infection and lost their HBsAg without seroconversion to anti-HBsAb.

ELIGIBILITY:
Inclusion Criteria:

Chronic Hepatitis B infection group

* 18-80 year-old
* Compensated liver disease
* Chronic HBV infection with or without NUCs treatment
* History of HBsAg positive > 6 months
* HBsAg negative with qualitative Elecsys (Roche) twice at least 6 months apart
* HBsAb negative
* HBV DNA < 20 IU/mL

Healthy group

* Healthy person without history of HBV vaccination (HBsAg, anti-HBc and HBsAb negative)

Exclusion Criteria:

* History of previous HBV vaccination
* Anti-HCV and/or anti-HIV positive
* Decompensated cirrhosis
* History of previous malignancies
* History or currently receive immunotherapy, cytotoxic or immunosuppressive agents
* Patient with immunodeficiency disease
* Creatinine > 1.5 mg/dL
* Pregnancy or lactating woman
* Unable to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
HBsAb level at 4 weeks after complete vaccine injection | an average of 7 months
  HBsAb level more than 10 mIU/ml at 7 months

SECONDARY OUTCOMES:
HBsAb level at 6 months after complete vaccine injection | an average of 1 year
  HBsAb level more than 10 mIU/ml at 6 months
Adverse event from HBV vaccine | an average of 1 year
  Any adverse event from HBV vaccine by CTCAE v4.0
Factors associated with HBV vaccine response | an average of 1 year
  Factors associated with HBV vaccine response at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tawesak Tanwandee, Principal Investigator — Department of Medicine, Faculty of medicine Siriraj Hospital, Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Taheri H, Hasanjani Roushan MR, Soleimani Amiri MJ, Pouralijan M, Bijani A. Efficacy of Hepatitis B vaccine in those who lost Hepatitis B surface antigen during follow-up: Efficacy of HBV vaccine in those who lost HBsAg. Hepat Mon. 2011 Feb;11(2):119-22. PMID 22087128